CLINICAL TRIAL: NCT03554421
Title: Percutaneous Tibial Nerve Stimulation - PTNS: an Alternative Treatment Option for Chronic Therapy Resistant Anal Fissure
Brief Title: Percutaneous Tibial Nerve Stimulation - an Alternative Treatment Option for Chronic Therapy Resistant Anal Fissure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: user
Record Dates: First submitted 2018-05-31; First posted 2018-06-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Chronic Anal Fissure
Keywords: Key Words: Anal Fissure, tibial nerve stimulation

STUDY DESIGN:
Intervention Model Description: Only patients with chronic anal fissures treated
Masking Description: Treatment known to both investigator and patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Posterior tibial nerve stimulation (Experimental): Percutaneous tibial nerve stimulation. Stimulation av posterior tibial nerve via neuromodulator for 30 minutes. 10 sessions
  Interventions: Procedure: Percutaneous tibial nerve stimulation

INTERVENTIONS:
Procedure: Percutaneous tibial nerve stimulation — A 20Hz electrical current is given via an electrode inserted through the skin over the posterior tibial nerve above the medial malleolus of the foot and the nerve is stimulated until a motor reflex of the big toe is acheived. Treatment is then continued for 30 minutes at this level. The treatment is then repeated for a total of 10 sessions within a 2 week period.

SUMMARY:
At a tertiary referral centre, 10 patients (4 male and 6 female; mean age 49.8 years) were given neuromodulation via the posterior tibial nerve to the sacral nerve for 30 min on 10 consecutive days. All patients had failed conventional medical treatment. The visual analogue scale (VAS), St. Marks score, Wexner's constipation score, Brief Pain Inventory (BPI - SF), bleeding and mucosal healing were evaluated before treatment, at termination, after 3 months and then yearly during three years.

DETAILED DESCRIPTION:
Between October 2013 and January 2014, 10 patients diagnosed with chronic anal fissure at the Pelvic Floor Centre - University Hospital of Malmo, Sweden were treated with percutaneous tibial nerve stimulation. Ethical clearance to use the results in a scientific setting was obtained from the ethics committee of the University of Lund, Sweden (Dnr 2016/998). Pre-treatment evaluation included detailed medical history and anorectal examination. All patients presented with pain and/or bleeding and the presence of a chronic anal fissure was confirmed by clinical examination.

Patients were included in the study if they were older than 18 years and had symptoms of chronic anal fissure for at least 6 months. All patients must have been on high fiber diet and stool softeners and in addition failed all conservative pharmacological treatment with topical application of anaesthetic creams, muscle relaxants (nitroglycerin or diltiazem) and/or botulinum toxin injection. We excluded patients with pregnancy, pacemaker device, low molecular heparin or warfarin treatment, neurological disease, inflammatory bowel disease and radiation proctitis. The Visual Analog Scale (VAS), St. Marks Incontinence Score, Wexner´s Constipation Score, Brief Pain Inventory - Short form (BPI-SF), symptom relief, bleeding and mucosal fissure healing were evaluated before and after treatment. VAS and BPI-SF were used to measure subjective pain characteristics and symptoms of patients at baseline, after two weeks (end of treatment), three months and then after one, two and three years. St. Marks Score and Wexner´s Constipation Score were evaluated in the same way though only up to one year after completion of treatment. The patients were given percutaneous tibial nerve stimulation after obtaining informed consent. The procedure was performed by two experienced pelvic floor therapists. Patients retained their high fiber diet and stool softeners during the procedure. Percutaneous tibial nerve stimulation was performed by using the Urgent PC Neuromodulation System ® (Uroplasty, Holland) on an outpatient basis. A stimulator provides electrical current with a fixed pulse frequency of 20Hz, pulse width 200 µ seconds and current setting between 0.5 and 9 mA (amplitude). A surface electrode was placed at the medial arch of the midfoot and a needle electrode was inserted through the skin posterior to the medial malleolus and advanced towards the posterior tibial nerve. Stimulation was gradually increased until a tingling sensation was perceived in the foot, or a motor flexor response was observed at the big toe. All patients received the treatment for 30 minutes 5 days a week, during 2 consecutive weeks. The clinical state of the fissure was evaluated before and after the last treatment session as well at three months and one year (though at the 3 month follow up one patient declined clinical examination since he felt completely symptom free). The fissure wound was characterized as not healed, partially healed when the healing process was visible but not totally complete and healed when no sign of the fissure was visible. At two and three years all patients were contacted by phone, and those who had symptoms where chronic anal fissure could not be ruled out underwent a clinical examination.

Statistical analyses:

The clinical outcome i.e. none healed, partially or totally healed fissure was analysed in relation to VAS, mean of St. Marks Incontinence Score and sum of Wexners's Constipation Score. These questions were chosen due to their clinical importance and high response rate. All analyses were calculated with descriptive statistics due to the few amount of patients. All analyses were performed with SPSS 22.

ELIGIBILITY:
Inclusion Criteria:

* 1. Chronic anal fissure for at least 6 months. 2. Above 18 years old. 3. Failed all previous conservative therapy. 4. On high fibre diet.

Exclusion Criteria:

* 1.Pregnancy 2. Pacemaker device. 3. Blood thinners - Heparin or Warfarin 4. Neurological disease 5. Inflammatory bowel disease 6. Radiation proctitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2014-02-11 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Rate of wound healing by clinical examination | 3 years
  Wound healing rate was assessed by visual Clinical examination of the wound taking into consideration the presence or absence of inflammation or epithelialization.
  The clinical state of the fissure wound was assessed in the scale of : not healed (more than 50% of wound visible), partially healed (more than 50% the healing process was visible but not totally complete) and healed when no sign of the active fissure or inflammation was visible and wound was completely epithilialized.

SECONDARY OUTCOMES:
Pain Intensity assessed by Visual Analogue Scale (VAS) | 3 years
  The severity and duration of pain was assessed by the Visual Analogue Scale where patients rated severity of pain om a 10 centimeter scale, ranging from 0 to 10. One end represents the lowest intensity of pain (0) and the other end of the scale representing the worst imaginable pain (10). The patient gives their indication with a pen mark on the line corresponding to the present pain level. Method of assessment is by interview.
Pain Inventory as assessed by Brief Pain Inventory (BPI-SF) | 3 years
  The pain inventory assesses the severity of pain and its impact on daily function, location of pain, pain medications and pain relief in the past 24 hours. Pain items monitored are: worst pain in last 24 hours, least pain in last 24 hours, pain on average, pain right now. Interference items assessed are: general activity, mood, normal work (including housework), relations with other people, sleep and enjoyment of Life.The scoring system is scaled from 0 to 10. The highest value correlating to worst pain possible or most interference in factors assessed. Pain relief after medication or treatment is assessed in percentiles from 0 % (least pain relief) to 100% (complete pain relief). The arithmetic mean of the four severity items can be used as measures of pain severity. The arithmetic mean of the seven interference items can be used as the measure of pain interference. Method of assessment is by self report or interview. Time required is about 5 minutes.
Bleeding of fissure wound as assessed by patient | 3 years
  Patients answered questionnaires by interview about the presence or absence of bleeding. They had to score a YES for bleeding and a NO for no bleeding
Bowel control as assessed by St. Marks Incontinence Score | 1 year
  The patients subjective perception of bowel control and incontinence for solid, liquid or gas is scored in a questionnaire between 0 and 4, where the highest score is equivalent to worst symptoms. The usage of constipatory medicines or pads is scored as 0 (No usage) or 2 (for Yes). The lack of ability to defer defecation for 15 minutes is scored as 0 (for No) and 4 (for Yes). The total score reflects the level of bowel Control, where 0 is complete continence and 24 equals complete incontinence.
Bowel movements assessed by Constipation Score | 1 year
  A constipation score with a scale of 0 to 4 for seven factors measured and a scale of 0 to 2 for assistance for evacuation. Total minimum score is 0 and maximum score of 30 indicating worst possible condition. Factors measured are; frequency of bowel movements, difficulty/painful evacuation effort, completeness/feeling of incomplete evacuation, pain (abdominal),time per evacuation, type of assistance, failure/unsuccessful attempts for evacuation per 24 hours, duration of constipation. Method of assessment by self report or interview.

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Jeppsson, Professor, Study Chair — Region Skane

IPD SHARING:
Plan to Share IPD: No
Nothing planned.